CLINICAL TRIAL: NCT02412592
Title: Sustained Viral Response and Clincal Relapse in Chronic Hepatitis B Patients Who Achieved HBeAg Seroncongversion by Interferon Therapy
Brief Title: Sustained Viral Response in Chronic Hepatitis B Patients Who Achieved HBeAg Seroncongversion After Interferon Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY009
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: HBeAg positive; interferon; peginterferon; HBeAg seroconversion; sustained viral response; relapse
MeSH Terms: conditions — Hepatitis B, Chronic; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic hepatitis B (CHB) is a serious liver disease worldwide, and the leading cause of cirrhosis and hepatocellular carcinoma (HCC). HBeAg seroconversion is considered to be the satisfied endpoint of antiviral therapy in HBeAg-positive chronic hepatitis B patients. However, HBV reaction, even reverse back to HBeAg positive and clinical relapse could occur in some patients who achieved HBeAg seronconversion by interferon treatment. In this study, the long-term efficacy of interferon therapy in HBeAg positive patients achieved HBeAg seronconversion after interferon treatment and the factors associated with viral and clinical relapse will be observed.

DETAILED DESCRIPTION:
HBeAg positive chronic hepatitis B patients achieved HBeAg seronconversion by interferon treatment will be enrolled and observed for 156 weeks. Serum HBV DNA, HBsAg, anti-HBs, HBeAg, and anti-HBe will be measured every 3 months during the observation period, liver function tests were performed every 3 months also. The liver ultrasonic examination would be taken every 3-6 months. The primary endpoint is sustained viral response, and secondary endpoints is HBV DNA reaction and clinical relapse defined as virla relapse with abnormal ALT during observation period.

ELIGIBILITY:
Inclusion Criteria:

* patients who achieved HBeAg seroconversion by interferon treatment.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population in this study were composed of HBeAg positive chronic hepatitis B patients achieved HBeAg seroconversion by interferon treatment, and serum HBsAg, anti-HBs, HBeAg, anti-HBe, and HBV DNA would be tested every 3 months for 156 weeks after finished treatment. The sustained viral response defined HBV DNA mantaining undetectable would be evalued during the observation period.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
sustained viral response | 156 weeks
  The serum HBV DNA load and HBeAg level will be tested every 3 month for 156 weeks after completed treatment in patients who achieved HBeAg seroconversion by interferon treatment. The rate of sustained viral response defined HBV DNA maintaining undetectable during observation period will be evaluated.

SECONDARY OUTCOMES:
HBV DNA reaction | 156 weeks
  HBV DNA reaction was defined as HBV DNA load reverse back to detectable during observation period.
clinical relapse | 156 weeks
  clinical relapse is defined as virla relapse with abnormal ALT during observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Yao Xie, Beijing, Beijing Municipality, China